CLINICAL TRIAL: NCT00828113
Title: Long-term Varenicline Treatment for Smoking Cessation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-2008-0149
Record Dates: First submitted 2009-01-21; First posted 2009-01-23 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Smoking
Keywords: smoking; relapse; withdrawal
MeSH Terms: conditions — Smoking; Recurrence | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended treatment (Experimental): 52-week varenicline therapy + individual smoking cessation counseling
  Interventions: Drug: varenicline; Behavioral: Individual smoking cessation counseling
- Standard treatment (Active Comparator): 13 weeks of varenicline therapy + individual smoking cessation counseling
  Interventions: Drug: varenicline; Behavioral: Individual smoking cessation counseling

INTERVENTIONS:
Drug: varenicline — Extension of 1 mg twice daily treatment to 52 weeks
Drug: varenicline — Double-blind switch to placebo after 12 weeks of open-label therapy
Behavioral: Individual smoking cessation counseling — Brief (<10 minutes) smoking cessation counseling delivered at clinic visits

SUMMARY:
This is a clinical study of the efficacy and safety of up to 52 weeks of varenicline therapy in conjunction with individual counseling for smoking cessation. Adult volunteers in generally good health, smoking 5 or more cigarettes per day, will receive 13 weeks of open-label varenicline therapy. At 12 weeks after their target quit date, they will be assigned in a random, double-blind manner to either 40 additional weeks of varenicline or placebo. It is hypothesized that biochemically-confirmed abstinence rates will be higher for the varenicline group at 52 weeks. Participants will be followed for an additional 26 weeks post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* daily smoker
* 5+ cigarettes per day for at least one year
* expired carbon monoxide level of 5+ ppm

Exclusion Criteria:

* current use of smoking cessation pharmacotherapies
* current or history of psychotic disorder
* current major depressive disorder
* history of suicidal ideation in the previous 3 months
* unstable medical condition
* pregnant, nursing, or planning to become pregnant
* planning to move from study area within 18 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Center for Tobacco Research and Intervention, Madison, Wisconsin
  - Center for Tobacco Research and Intervention, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Extended Treatment | Standard Treatment
Started | 50 | 51
Completed | 20 | 20
Not Completed | 30 | 31
Not completed — Withdrawal by Subject | 27 | 26
Not completed — Lost to Follow-up | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended Treatment | Standard Treatment | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 51 | 101
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (11.6) | 43.2 (12.4) | 42.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 29 | 29 | 58
Region of Enrollment [Number; unit: participants]
  United States | 50 | 51 | 101

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Not Smoking in the Previous 7 Days, Confirmed by Expired Carbon Monoxide Reading < 10 Parts Per Million at Week 52
Description: Self-report of no smoking (not even a puff) in the previous seven days confirmed by an expired carbon monoxide reading of < 10 parts per million as assessed at Week 52
Time Frame: 7-day point prevalence
Population: Participants randomized at 12 weeks who continued in the study to Week 52 and provided CO-verified smoking status.
Measure: Number; unit: participants
Arm/Group | Extended Treatment | Standard Treatment
Number analyzed (Participants) | 33 | 34
participants | 10 | 11

ADVERSE EVENTS:
Description: Number of participants at risk based upon those available to be randomized at Week 12
Arm/Group | Extended Treatment | Standard Treatment
Serious Adverse Events (participants affected / at risk) | 1/33 | 1/34
Other Adverse Events (participants affected / at risk) | 13/33 | 12/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Extended Treatment (N=33) | Standard Treatment (N=34)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 0 | 1
Bladder Surgery (Renal and urinary disorders) | 1 | 0 — Occurred two months into nontreatment follow-up phase
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Extended Treatment (N=33) | Standard Treatment (N=34)
Nausea (Gastrointestinal disorders) | 2 | 0
General Disorders NOS (General disorders) | 1 | 3
Upper Respiratory Tract Disorder (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Respiratory NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Metabolism NOS (Metabolism and nutrition disorders) | 2 | 0
Infection NOS (Infections and infestations) | 3 | 2
Musculoskeletal NOS (Musculoskeletal and connective tissue disorders) | 3 | 4
Hypertension (Vascular disorders) | 2 | 4
Injuries (Injury, poisoning and procedural complications) | 3 | 1

LIMITATIONS AND CAVEATS:
Feasibility study with limited statistical power at baseline compounded by a significant rate of attrition during the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less